CLINICAL TRIAL: NCT03151707
Title: The Effects of Nicotinamide Riboside Supplementation on Nicotinamide Adenine Dinucleotide (NAD+/NADH) Ratio and Bioenergetics
Brief Title: The Effects of Nicotinamide Riboside Supplementation on Brain NAD+/NADH Ratio and Bioenergetics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding and appropriate staff
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Dost Ongur, Chief of Psychotic Disorders Division at McLean Hospital and Associate Professor in Psychiatry at Harvard Medical School, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000006
Record Dates: First submitted 2017-05-04; First posted 2017-05-12 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nicotinamide riboside 2g/day (Experimental): Participants will receive NR at a dose of 2g/day
  Interventions: Drug: Nicotinamide Riboside

INTERVENTIONS:
Drug: Nicotinamide Riboside — Nicotinamide riboside 2g/day for a 2 week duration

SUMMARY:
The primary aim of this study is to investigate the effects of exogenously administered nicotinamide riboside (NR) on brain NAD+/NADH ratio and bioenergetics functions in healthy individuals using phosphorus magnetic resonance spectroscopy (31P MRS) imaging.

The secondary aims are to investigate the change in brain PCr/ATP and creatine kinase enzyme rate after NR use. In addition, NAD+/NADH ratio, PCr/ATP and CK enzyme rate will be measured in the calf muscle, as secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 year-old
2. Male or female
3. Without psychiatric diagnosis according to a structured psychiatric interview (Structured Clinical Interview for DSM-V Axis I Disorders (SCID))
4. Without history of a psychotic disorder and/or mood disorder among parents, siblings, or children, as obtained via self-report only.

Exclusion Criteria:

1. Significant medical or neurological illness.
2. Diagnosis diabetes mellitus (DM), uncontrolled hypertension (HTN), severe hypotension, coronary artery disease (CAD), metabolic syndrome, glaucoma, liver impairment, decreased renal function, respiratory disorders, uncontrolled peptic ulcer disease.
3. Taking any other medications, including over the counter supplements with the exception of oral contraceptives for women
4. Pregnancy. Females of child-bearing age must be using an effective contraceptive method.
5. History of smoking, substance abuse or dependence.
6. Contraindication to MR scan (claustrophobia, cardiac pacemakers, metal clips and stents on blood vessels, artificial heart valves, artificial arms, hands, legs, etc., brain stimulator devices, implanted drug pumps, ear implants, eye implants or known metal fragments in eyes, exposure to shrapnel or metal filings, other metallic surgical hardware in vital areas, certain tattoos with metallic ink, certain transdermal patches, metal- containing intrauterine devices)
7. Medical condition that would prevent blood draws, including current anti-coagulant or anti-aggregant therapy, tendency for abnormal scarring (e.g. keloids).
8. Difficulty in swallowing capsules.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dost Ongur, MD PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotinamide Riboside 2g/Day
Started | 11
Completed | 5
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Nicotinamide Riboside 2g/Day
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
NAD+/NADH Ratio [Mean (Standard Deviation); unit: Ratio] — NAD+/NADH ratio is calculated by first quantifying NAD+ and NADH separately in MR Spectroscopy data and then obtaining a simple ratio of the 2 measures.
  There is a normative ratio in healthy brain and deviations from this ratio in either direction can be a sign of pathology. Population: Early termination led to data not being available from all participants
  Ratio
    number analyzed (Participants) | 4
    (all) | 3.75 (0.47)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of Treatment in Brain NAD+/NADH Ratio
Description: Change from baseline to the end of treatment in brain NAD+/NADH ratio as measured by in vivo 31P magnetic resonance spectroscopy
  The NAD+/NADH ratio is calculated by first quantifying NAD+ and NADH separately in the data and then obtaining a simple ratio. There is a normative NAD+/NADH ratio range in healthy brain and deviations from this level in either direction can be a sign of pathology.
Time Frame: Baseline and after 15 days of supplement use
Population: Early termination led to small number of subjects analyzed
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Nicotinamide Riboside 2g/Day
Number analyzed (Participants) | 4
Ratio | 0.198 (0.025)

2. Secondary Outcome: Change From Baseline to the End of Treatment in Brain Phosphocreatine (PCr) to Adenosine Triphosphate (ATP) Ratio (PCr/ATP)
Description: Change from baseline to the end of treatment in brain phosphocreatine (PCr) to adenosine triphosphate (ATP) ratio (PCr/ATP) as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: Baseline and after 15 days of supplement use
Population: No data were collected/analyzed for this measure.
Arm/Group | Nicotinamide Riboside 2g/Day
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline to the End of Treatment in Brain Creatine Kinase (CK) Enzyme Rate
Description: Change from baseline to the end of treatment in creatine kinase (CK) enzyme rate as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: Baseline and after 15 days of supplement use
Population: No data were collected/analyzed for this measure.
Arm/Group | Nicotinamide Riboside 2g/Day
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline to the End of Treatment in Muscle NAD+/NADH Ratio
Description: Change from baseline to the end of treatment in calf muscle NAD+/NADH ratio as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: Baseline and after 15 days of supplement use
Population: No data were collected/analyzed for this measure.
Arm/Group | Nicotinamide Riboside 2g/Day
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline to the End of Treatment in Muscle Phosphocreatine (PCr) to Adenosine Triphosphate (ATP) Ratio (PCr/ATP)
Description: Change from baseline to the end of treatment in calf muscle phosphocreatine (PCr) to adenosine triphosphate (ATP) ratio (PCr/ATP) as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: Baseline and after 15 days of supplement use
Population: No data were collected/analyzed for this measure.
Arm/Group | Nicotinamide Riboside 2g/Day
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline to the End of Treatment in Muscle Creatine Kinase (CK) Enzyme Rate
Description: Change from baseline to the end of treatment in calf muscle creatine kinase (CK) enzyme rate as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: Baseline and after 15 days of supplement use
Population: No data were collected/analyzed for this measure.
Arm/Group | Nicotinamide Riboside 2g/Day
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 15 days
Arm/Group | Nicotinamide Riboside 2g/Day
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide Riboside 2g/Day (N=11)
Mild Nausea (Gastrointestinal disorders) | 1 (1)
Mild stomach pain (Gastrointestinal disorders) | 1 (1)
Bruising at blood draw site (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT03151707/Prot_001.pdf